CLINICAL TRIAL: NCT06131437
Title: Efficacy and Safety of Cagrilintide 2.4 mg s.c. in Combination With Semaglutide 2.4 mg s.c. (CagriSema s.c. 2.4 mg/2.4 mg) Once-weekly Compared to Tirzepatide 15 mg s.c. Once-weekly in Participants With Obesity
Brief Title: A Research Study to See How Well CagriSema Compared to Tirzepatide Helps People With Obesity Lose Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-7832; U1111-1292-4835 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide; Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema 2.4 mg/2.4 mg (Experimental): Participants will receive 2.4 mg cagrilintide and 2.4 mg semaglutide subcutaneously once-weekly (dose escalation period of 16 weeks) for up to 84 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Tirzepatide 15 mg (Active Comparator): Participants will receive 15 mg tirzepatide subcutaneously once-weekly (dose escalation period of 20 weeks) for up to 84 weeks.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Cagrilintide — Cagrilintide will be administered subcutaneously.
  Arms: CagriSema 2.4 mg/2.4 mg
Drug: Semaglutide — Semaglutide will be administered subcutaneously.
  Arms: CagriSema 2.4 mg/2.4 mg
Drug: Tirzepatide — Tirzepatide will be administered subcutaneously.
  Arms: Tirzepatide 15 mg

SUMMARY:
This study will look at how well CagriSema compared to Tirzepatide helps people lower their body weight. CagriSema is a new investigational medicine developed by Novo Nordisk that combines Cagrilintide and Semaglutide. CagriSema is not yet being prescribed by doctors. Participant will get injections once a week throughout the treatment period. Participant will inject the study medicine under the skin with a pen injector in the thigh, stomach, or upper arm. After a first low dose, the study medicine will be gradually increased until reaching the planned dose (2.4 mg CagriSema or 15 mg Tirzepatide). The study will last for about one and a half year for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 years or above at the time of signing the informed consent
* Body mass index (BMI) of ≥ 30.0 kilogram per square meter (kg/m^2)

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) ≥ 6.5 % (48 millimoles per mole [mmol/mol]) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 809 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
To confirm non-inferiority of CagriSema versus tirzepatide: Relative change in body weight | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage (%).

SECONDARY OUTCOMES:
To confirm superiority of CagriSema versus tirzepatide: Relative change in body weight | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage (%).
Achievement of greater than or equal to (≥) 25% weight reduction | From baseline (week 0) to end of treatment (week 84)
  Count of participants.
Achievement of ≥ 30% weight reduction | From baseline (week 0) to end of treatment (week 84)
  Count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 84)
  Measured in centimeter (cm).
Change in systolic blood pressure (SBP) | From baseline (week 0) to end of treatment (week 84)
  Measured in millimeter of mercury (mmHg).
Change in diastolic blood pressure (DBP) | From baseline (week 0) to end of treatment (week 84)
  Measured in mmHg.
Relative change in lipids: Total cholesterol | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Relative change in lipids: High-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Relative change in lipids: Non-HDL cholesterol | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Relative change in lipids: Low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Relative change in lipids: Very low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Relative change in lipids: Triglycerides | From baseline (week 0) to end of treatment (week 84)
  Measured in percentage.
Number of Treatment-emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 90)
  Count of events.
Number of Treatment Emergent Serious adverse events (TESAEs) | From baseline (week 0) to end of study (week 90)
  Count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (46):
- United States (46):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Chambliss Clinical Trials LLC, Montgomery, Alabama
  - FDRC, Costa Mesa, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Univ of Colorado at Denver, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Northeast Research Institute, Fleming Island, Florida
  - Jacksonville Ctr For Clin Res, Jacksonville, Florida
  - South Broward Research LLC, Miramar, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Endeavor Health, Skokie, Illinois
  - Evanston Premier Hlthcr Res, Skokie, Illinois
  - Midwest Inst For Clin Res, Indianapolis, Indiana
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Comprehensive Weight Ctrl Prog, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Accellacare_NC, Raleigh, North Carolina
  - Accellacare, Wilmington, North Carolina
  - New Venture Medical Research, Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - The University of Penn Center, Philadelphia, Pennsylvania
  - Clinical Res Collaborative, Cumberland, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina
  - Coastal Carolina Res Ctr, North Charleston, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Elligo Clin Res Centre, Austin, Texas
  - UT Health University of Texas, Bellaire, Texas
  - Baylr Sctt White Rs Inst, Endo, Dallas, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - UT Southwestern Medical Center-CRU, Dallas, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Health Res of Hampton Roads, Newport News, Virginia
  - National Clin Res Inc., Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Capital Clin Res Ctr,LLC, Olympia, Washington
  - Rainier Clin Res Ctr Inc, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com